CLINICAL TRIAL: NCT04929223
Title: A Phase I/Ib Global, Multicenter, Open-label Umbrella Study Evaluating the Safety and Efficacy of Targeted Therapies in Subpopulations of Patients With Metastatic Colorectal Cancer (INTRINSIC)
Brief Title: A Study Evaluating the Safety and Efficacy of Targeted Therapies in Subpopulations of Patients With Metastatic Colorectal Cancer (INTRINSIC)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO42758; 2021-001207-33 (EudraCT Number); 2023-505163-37-00 (Other: CTIS (EU))
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: KRAS G12C
MeSH Terms: conditions — Colorectal Neoplasms | interventions — inavolisib; Bevacizumab; Cetuximab; atezolizumab; Tiragolumab; SY-5609; Folfox protocol; IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Inavolisib + Cetuximab (Experimental): Participants will receive 9 milligrams (mg) of inavolisib by mouth once daily (QD) on Days 8-28 of Cycle 1, then QD on Days 1-28 from Cycle 2 onwards (1 cycle=28 days).
  Participants will also receive cetuximab intravenous (IV) infusion 400 mg/m2 body surface area on Day 1 of Cycle 1. All subsequent weekly (QW) doses will be 250 mg/m2 each. This arm is closed.
  Interventions: Drug: Inavolisib; Drug: Cetuximab; Diagnostic Test: FoundationOne®Liquid CDx
- Inavolisib + Bevacizumab (Experimental): Participants will receive 9 mg of inavolisib by mouth QD combined with bevacizumab 15 milligram/kilogram (mg/kg) IV once every three weeks (Q3W) on Day 1 of each cycle (1 cycle=21 days). This arm is closed.
  Interventions: Drug: Inavolisib; Drug: Bevacizumab; Diagnostic Test: FoundationOne®Liquid CDx
- Atezolizumab + Tiragolumab + Bevacizumab (Experimental): Participants in this randomized cohort will receive 1200 mg of atezolizumab by IV infusion on Day 1 of each cycle, combined with tiragolumab at a dose of 600 mg IV infusion on Day 1 of each cycle and bevacizumab IV infusion at a dose of 15 mg/kg on Day 1 of each cycle. (Cycle length=21 days) This arm is active, and not recruiting participants.
  Interventions: Drug: Bevacizumab; Drug: Atezolizumab; Drug: Tiragolumab; Diagnostic Test: FoundationOne®Liquid CDx
- Atezolizumab + Tiragolumab (Experimental): Participants in this randomized cohort will receive 1200 mg of atezolizumab by IV infusion on Day 1 of each cycle combined with tiragolumab 600 mg IV infusion on Day 1 of each cycle. (Cycle length=21 days) This arm is active, and not recruiting participants.
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab; Diagnostic Test: FoundationOne®Liquid CDx
- Atezolizumab + SY-5609 (Experimental): Participants will receive 1680 mg of atezolizumab by IV infusion on Day 1 of each cycle Q4W in repeated 28-day cycles combined with SY-5609 at a dose of 3, 4, 5, 6, 7 or 10 mg by mouth for 7 days, followed by 7 days off. (Cycle length=28 days) This arm is closed.
  Interventions: Drug: Atezolizumab; Drug: SY-5609; Diagnostic Test: FoundationOne®Liquid CDx
- Divarasib + Cetuximab + FOLFOX (Experimental): Participants will receive cetuximab IV 500 mg/m2 body surface area on Days 1 and 15 and FOLFOX on Days 1 and 15 with divarasib PO QD on Days 1-28. (Cycle length=28 days) This arm is recruiting participants.
  Interventions: Drug: Cetuximab; Drug: Divarasib; Drug: FOLFOX; Diagnostic Test: FoundationOne®Liquid CDx
- Divarasib + Cetuximab (Experimental): Participants will receive cetuximab IV 500 mg/m2 body surface area on Days 1 and 15 with divarasib PO QD on Days 1-28. (Cycle length=28 days) This arm is active, and not recruiting participants.
  Interventions: Drug: Cetuximab; Drug: Divarasib; Diagnostic Test: FoundationOne®Liquid CDx
- Divarasib + Cetuximab + FOLFIRI (Experimental): Participants will receive cetuximab IV 500 mg/m2 body surface area on Days 1 and 15 and FOLFIRI on Days 1 and 15 with divarasib PO QD on Days 1-28. (Cycle length=28 days) This arm is active, and not recruiting participants.
  Interventions: Drug: Cetuximab; Drug: Divarasib; Drug: FOLFIRI; Diagnostic Test: FoundationOne®Liquid CDx
- Divarasib + Bevacizumab + FOLFOX (Experimental): Participants will receive Bevacizumab 5 mg/kg by IV infusion on Days 1 and 15 and FOLFOX on Days 1 and 15 with Divarasib PO QD on Days 1-28. (Cycle length=28 days) This arm is recruiting participants.
  Interventions: Drug: Bevacizumab; Drug: Divarasib; Drug: FOLFOX; Diagnostic Test: FoundationOne®Liquid CDx
- Divarasib + Bevacizumab + FOLFIRI (Experimental): Participants will receive Bevacizumab 5 mg/kg by IV infusion on Days 1 and 15 and FOLFIRI on Days 1 and 15 with Divarasib PO QD on Days 1-28. (Cycle length=28 days) This arm is recruiting participants.
  Interventions: Drug: Bevacizumab; Drug: Divarasib; Drug: FOLFIRI; Diagnostic Test: FoundationOne®Liquid CDx

INTERVENTIONS:
Drug: Inavolisib — Inavolisib will be administered orally as per schedule specified in the respective arms.
  Arms: Inavolisib + Bevacizumab; Inavolisib + Cetuximab
Drug: Bevacizumab — Bevacizumab IV will be administered as per schedule specified in the respective arm.
  Other Names: Avastin
  Arms: Atezolizumab + Tiragolumab + Bevacizumab; Divarasib + Bevacizumab + FOLFIRI; Divarasib + Bevacizumab + FOLFOX; Inavolisib + Bevacizumab
Drug: Cetuximab — Cetuximab IV will be administered as per schedule specified in the respective arm.
  Arms: Divarasib + Cetuximab; Divarasib + Cetuximab + FOLFIRI; Divarasib + Cetuximab + FOLFOX; Inavolisib + Cetuximab
Drug: Atezolizumab — Atezolizumab IV infusion will be administered as per schedule specified in the respective arm.
  Other Names: Tecentriq
  Arms: Atezolizumab + SY-5609; Atezolizumab + Tiragolumab; Atezolizumab + Tiragolumab + Bevacizumab
Drug: Tiragolumab — Tiragolumab IV infusion will be administered as per schedule specified in the respective arm.
  Arms: Atezolizumab + Tiragolumab; Atezolizumab + Tiragolumab + Bevacizumab
Drug: SY-5609 — SY-5609 will be administered by mouth as per schedule specified in the respective arm.
  Arms: Atezolizumab + SY-5609
Drug: Divarasib — Divarasib will be administered orally as per schedule specified in the respective arms.
  Other Names: GDC-6036
  Arms: Divarasib + Bevacizumab + FOLFIRI; Divarasib + Bevacizumab + FOLFOX; Divarasib + Cetuximab; Divarasib + Cetuximab + FOLFIRI; Divarasib + Cetuximab + FOLFOX
Drug: FOLFOX — FOLFOX (5-fluorouracil, leucovorin, oxaliplatin) IV will be administered as per schedule specified in the respective arm.
  Arms: Divarasib + Bevacizumab + FOLFOX; Divarasib + Cetuximab + FOLFOX
Drug: FOLFIRI — FOLFIRI (leucovorin, 5-fluorouracil, irinotecan) IV will be administered as per schedule specified in the respective arm.
  Arms: Divarasib + Bevacizumab + FOLFIRI; Divarasib + Cetuximab + FOLFIRI
Diagnostic Test: FoundationOne®Liquid CDx — FoundationOne®Liquid CDx is used to identify presence of genomic alterations for participant cohort assignment.

SUMMARY:
This open-label, exploratory study is designed to evaluate the safety and efficacy of targeted therapies or immunotherapy as single agents or combinations, in participants with metastatic colorectal cancer (mCRC) whose tumors are biomarker positive as per treatment arm-specific definition. Eligible participants with mCRC will be enrolled into specific treatment arms based on their biomarker assay results.

ELIGIBILITY:
Inclusion Criteria

* Signed cohort-specific Informed Consent Form
* Age >= 18 years at time of signing Informed Consent Form
* Biomarker eligibility as determined by:

  * A validated test approved by local health authorities for detection of the specified biomarkers/mutations.
  * A validated test performed at a College of American Pathologists/clinical laboratory improvement amendments (CAP/CLIA) -certified or equivalently accredited diagnostic laboratory using a validated test for detection of the specified biomarkers.
  * Prior test results completed before signing cohort-specific Informed Consent Form or local test results generated prior to or during screening, and availability of a full report of the testing results OR
  * Blood-based FoundationOne Liquid CDx biomarker eligibility test result generated prior to or during screening or, in case of re-enrollment after treatment discontinuation, prior to starting a new anti-cancer therapy.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of <= 1
* Life expectancy >= 3 months, as determined by the investigator
* Histologically confirmed adenocarcinoma originating from the colon or rectum
* Metastatic disease
* Prior therapies for metastatic disease
* Ability to comply with the study protocol, in the investigators judgment
* Measurable disease (at least one target lesion) according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1)
* Baseline tumor tissue samples will be collected from all participants for exploratory biomarker research
* Adequate hematologic and organ function within 14 days prior to initiation of study treatment
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures
* For men: agreement to remain abstinent or use contraceptive measures, and agreement to refrain from donating sperm

Exclusion Criteria

* Current participation or enrollment in another interventional clinical trial. Participants who are participating in the follow-up period of an interventional clinical trial are eligible for the study.
* Any systemic anti-cancer treatment within 2 weeks or 5 half-lives (whichever is shorter) prior to start of study treatment
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Pregnant or breastfeeding, or intending to become pregnant during the study
* History of or concurrent serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study or confounds the ability to interpret data from the study
* Severe infection within 4 weeks prior to initiation of study treatment or any active infection that, in the opinion of the investigator, could impact patient safety
* Incomplete recovery from any surgery prior to the start of study treatment that would interfere with the determination of safety or efficacy of study treatment
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)
* Uncontrolled tumor-related pain
* Uncontrolled or symptomatic hypercalcemia
* Clinically significant and active liver disease
* Negative HIV test at screening, with the following exception: Participants with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy for at least 4 weeks, have a CD4 count greater than or equal to 200/uL, have an undetectable viral load, and have not had a history of opportunistic infection attributable to AIDS within the last 12 months.
* Symptomatic, untreated, or actively progressing CNS metastases
* History of leptomeningeal disease or carcinomatous meningitis
* History of malignancy other than CRC within 2 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death
* Any other disease, unresolved toxicity from prior therapy, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the participant at high risk from treatment complications
* Requirement for treatment with any medicinal product that contraindicates the use of any of the study treatments, may interfere with the planned treatment, affects participant compliance, or puts the patient at higher risk for treatment-related complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2030-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Approximately 84 months
  Defined as the proportion of participants with a complete response or partial response, as determined by the investigator according to RECIST v1.1

SECONDARY OUTCOMES:
Duration of Response | Approximately 84 months
  Defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1
Disease Control Rate | Approximately 84 months
  Defined as the proportion of participants with stable disease, or a complete or partial response, as determined by the investigator according to RECIST v1.1
Percentage of Participants with Adverse Events (AEs) | Approximately 84 months
  Percentage of participants with adverse events.
Plasma Concentrations of Divarasib | At pre-defined intervals from first administration of study drug up to approximately 84 months
  Plasma concentration of divarasib for divarasib + cetuximab + FOLFOX, divarasib + cetuximab, and divarasib + cetuximab+ FOLFIRI, Divarasib + Bevacizumab + FOLFOX, Divarasib + Bevacizumab + FOLFIRI treatment arms.
Recommended Dose of Divarasib in Combination with Bevacizumab and FOLFOX | Approximately 84 months
  Recommended dose of divarasib in combination with bevacizumab and FOLFOX based on the totality of safety, efficacy and PK data.
Recommended Dose of Divarasib in Combination with Bevacizumab and FOLFIRI | Approximately 84 months
  Recommended dose of divarasib in combination with bevacizumab and FOLFIRI based on the totality of safety, efficacy and PK data.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (73):
- United States (30):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Mayo Clinic Arizona, Phoenix, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - cCare, Encinitas, California
  - USC Norris Cancer Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Stanford Cancer Center, Stanford, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Eastern Ct Hema/Onco Assoc, Norwich, Connecticut
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Mary Bird Perkins Cancer Ctr, Baton Rouge, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - New York Cancer & Blood Specialists - New Hyde Park, New Hyde Park, New York
  - New York Cancer and Blood Specialists-Central Park Hematology & Oncology, New York, New York
  - New York Cancer & Blood Specialists, Port Jefferson Station, New York
  - New York Cancer & Blood Specialists - Bronx, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Hematology Oncology Salem, Salem, Oregon
  - UPMC - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute / Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Lumi Research, Kingwood, Texas
  - Swedish Cancer Inst., Seattle, Washington
  - Medical Oncology Associates, Spokane, Washington
- Peter Maccallum Cancer Centre, Melbourne, Victoria, Australia
- Canada (3):
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
- Rigshospitalet, Onkologisk Klinik, København Ø, Denmark
- Germany (8):
  - Charité Universitätsmedizin Berlin, Berlin
  - Katholisches Klinikum Bochum gGmbH - St. Josef-Hospital, Bochum
  - Universitätsklinik Carl Gustav Carus der Technischen Universität Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Asklepios Klinik Altona, Hamburg
  - SLK-Kliniken Heilbronn GmbH;Klinik für Innere Medizin III, Heilbronn
  - Klinikum der Universität München, Campus Großhadern, München
  - Universitätsklinikum Ulm, Ulm
- Italy (5):
  - Università degli Studi della Campania Luigi Vanvitelli, Napoli, Campania
  - Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio
  - Irccs Istituto Nazionale Dei Tumori (Int), Milan, Lombardy
  - Azienda Socio Sanitaria Territoriale Niguarda (Ospedale Niguarda Ca' Granda), Milan, Lombardy
  - IRCCS Istituto Oncologico Veneto (IOV), Padua, Veneto
- Poland (3):
  - Szpital Uniwersytecki w Krakowie, Oddzia? Kliniczny Kliniki Onkologii, Krakow
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Narodowy Instytut Onkologii im. M. Sklodowskiej-Curie, Warsaw
- South Korea (7):
  - National Cancer Center, Goyang-si
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Seoul National University Bundang Hospital, Seongnam-si
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (4):
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - START Madrid-FJD, Hospital Fundacion Jimenez Diaz, Madrid
  - START Madrid. Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Clínico Universitario de Valencia, Valencia
- Taiwan (3):
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital, Zhongzheng Dist.
- United Kingdom (8):
  - Addenbrookes Hospital, Cambridge
  - Velindre Cancer Centre, Cardiff
  - Royal Free Hospital, London
  - Royal Marsden Hospital;Dept of Med-Onc, London
  - Sarah Cannon Research Institute, London
  - Imperial College Healthcare NHS Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: No